CLINICAL TRIAL: NCT07100288
Title: Anatomopathological Analysis of the Infundibulopelvic Ligament in Patients With Ovarian Cancer
Acronym: INFPELV
Status: Recruiting | Type: Observational
Sponsor: Complejo Hospitalario Universitario Insular Materno Infantil (Other)
Responsible Party: Principal Investigator, Beatriz Fatima Navarro Santana, GYNECOLOGIST ONCOLOGIST, Complejo Hospitalario Universitario Insular Materno Infantil
Other Study IDs: 2024-430-1
Record Dates: First submitted 2025-07-20; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Ovarian Cancer; Ovarian Cancer (OvCa); Ovarian Adenocarcinoma
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ovarian cancer patients
  Interventions: Other: resection of infundibulopelvic ligament

INTERVENTIONS:
Other: resection of infundibulopelvic ligament — Therefore, this study also aims to perform bilateral infundibulopelvic ligament resection (at least 8 cm in length) during surgery for ovarian cancer patients

SUMMARY:
Involvement of the infundibulopelvic ligament in ovarian cancer may be associated with decreased survival and related to paraaortic lymph node metastasis

ELIGIBILITY:
Inclusion Criteria:

* ◦ Patients with epithelial ovarian cancer, including high- and low-grade serous, high- and low-grade endometrioid, mucinous (expansile and infiltrative types), and carcinosarcoma.

  * FIGO 2014 stage IA-IVB.
  * Patients undergoing primary surgery or interval surgery after 3-4 or 6 cycles of chemtherapy
  * Patients with no residual disease after surgery.
  * Patients with ECOG performance status 0-1.

Exclusion Criteria:

* ◦ Patients without epithelial ovarian cancer.

  * Patients with ECOG 2-4.
  * Patients who do not consent to participate in the study.
  * Patients who did not undergo complete staging surgery (including hysterectomy, bilateral salpingo-oophorectomy, pelvic and para-aortic lymphadenectomy, and omentectomy) or with residual disease after cytoreductive surgery.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with FIGO stage IA-IVB epithelial ovarian cancer who undergoing surgery at our center.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-07-20 (Actual); Primary Completion 2030-07-20 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
metastasis in infundibulopelvic ligament | Through study completion, an average of 5 year
  To analyze the percentage of infundibulopelvic ligament involvement by cancer in patients with FIGO stage IA-IVB ovarian cancer.

SECONDARY OUTCOMES:
Presence of paraaortic lymph node metastasis | Through study completion, an average of 5 year
  Evaluation of histologically positive para-aortic lymph nodes in patients with metastasis in the infundibulopelvic ligament

OTHER OUTCOMES:
Disease Free Survival | 3 months, 6 months, 9 months, 12 months, 15 months, 18 months, 21 months, 24 months, 27 months, 30 months, 33 months, 36 months, 42 months, 48 months, 54 months, 60 months
  Impact of infundibulopelvic ligament involvement on Disease specific survival
Assessment of complications | during surgery, at hospital discharge, day 30
  Assessment of perioperative complications and site effects of infundibulopelvic ligament resection
Overall survival (OS) | 60 months
  Impact of infundibulopelvic ligament involvement on overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- Complejo Universitario Insular Materno Infantil de Las Palmas, Las Palmas de Gran Canaria, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tozzi R, Kohler C, Ferrara A, Schneider A. Laparoscopic treatment of early ovarian cancer: surgical and survival outcomes. Gynecol Oncol. 2004 Apr;93(1):199-203. doi: 10.1016/j.ygyno.2004.01.004. PMID 15047236
- [Background] Kleppe M, Kraima AC, Kruitwagen RF, Van Gorp T, Smit NN, van Munsteren JC, DeRuiter MC. Understanding Lymphatic Drainage Pathways of the Ovaries to Predict Sites for Sentinel Nodes in Ovarian Cancer. Int J Gynecol Cancer. 2015 Oct;25(8):1405-14. doi: 10.1097/IGC.0000000000000514. PMID 26397066
- [Background] Fennimore IA, Simon NL, Bills G, Dryfhout VL, Schniederjan AM. Extension of ovarian tissue into the infundibulopelvic ligament beyond visual margins. Gynecol Oncol. 2009 Jul;114(1):61-3. doi: 10.1016/j.ygyno.2009.03.006. Epub 2009 Apr 9. PMID 19361838
- Available data/document: preprint — https://www.researchsquare.com/article/rs-283444/v1